CLINICAL TRIAL: NCT04047225
Title: POSTOPERATIVE OPIOID-SPARING EFFECT OF INTRAOPERATIVE PAIN MONITORING USING THE ANALGESIA NOCICEPTIVE INDEX (ANI) DURING IDIOPATHIC SCOLIOSIS CORRECTION IN CHILDREN.
Acronym: OpiSpANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: APHP180604; 2019-A01388-49 (Other: ID-RCB)
Record Dates: First submitted 2019-08-05; First posted 2019-08-06 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2021-10

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Intervention Model Description: THE ANALGESIA NOCICEPTIVE INDEX (ANI)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia Nociceptive Index (ANI) (Experimental): Using ANI for guiding intraoperative opioid administration.
  Interventions: Device: THE ANALGESIA NOCICEPTIVE INDEX (ANI)
- No Analgesia Nociceptive Index (ANI) (No Intervention): Do not use ANI

INTERVENTIONS:
Device: THE ANALGESIA NOCICEPTIVE INDEX (ANI) — Utilisation of the ANI during the operation
  Other Names: THE ANALGESIA NOCICEPTIVE INDEX
  Arms: Analgesia Nociceptive Index (ANI)

SUMMARY:
Anaesthesia is often performed using a balanced technique by administering both opioids and anaesthetics agents. Intraoperative opioid administration is still relying on simple parameters such as heart rate and blood pressure variations. However, many studies in both adults and children have shown the poor accuracy of those parameters in predicting pain because of their sensibility to other intraoperative events such as depth of anaesthesia and volaemic variations. Consequently, intraoperative analgesia is still inadequately managed with periods of under dosage or over dosage of opioid agents. This has been hypothesized to cause postoperative hyperalgesia related to both intraoperative pain (in case of under dosage) or to opioid agents (in case of over dosage). The main resulting effect is an increase of postoperative opioid consumption and the inadequate postoperative rehabilitation because of adverse effects of opioids.

During the last decade, many pain-monitors have been investigated. Most of these devices are relying on the determination of the sympathetic-to the parasympathetic systems balance. Among those monitors, the Analgesia Nociceptive Index (ANI) quantifies the parasympathetic system. The ANI device can produce two parameters the instantaneous ANI (ANIi), derived from 60 seconds analysis and the mean ANI (ANIm) derived from 4 minutes analysis. Studies have shown the accuracy of ANIi to detect both experimental and clinical pain in various populations. Moreover, a recent randomized controlled trial during spine surgery in adults has found ANIi to decrease the intraoperative and postoperative opioid consumption when used intraoperatively for guiding the administration of opioid agents

DETAILED DESCRIPTION:
Anaesthesia is often performed using a balanced technique by administering both opioids and anaesthetics agents. Intraoperative opioid administration is still relying on simple parameters such as heart rate and blood pressure variations. However, many studies in both adults and children have shown the poor accuracy of those parameters in predicting pain because of their sensibility to other intraoperative events such as depth of anaesthesia and volaemic variations. Consequently, intraoperative analgesia is still inadequately managed with periods of under dosage or over dosage of opioid agents. This has been hypothesized to cause postoperative hyperalgesia related to both intraoperative pain (in case of under dosage) or to opioid agents (in case of over dosage). The main resulting effect is an increase of postoperative opioid consumption and the inadequate postoperative rehabilitation because of adverse effects of opioids.

During the last decade, many pain-monitors have been investigated. Most of these devices are relying on the determination of the sympathetic-to the parasympathetic systems balance. Among those monitors, the Analgesia Nociceptive Index (ANI) quantifies the parasympathetic system. The ANI device can produce two parameters the instantaneous ANI (ANIi), derived from 60 seconds analysis and the mean ANI (ANIm) derived from 4 minutes analysis. Studies have shown the accuracy of ANIi to detect both experimental and clinical pain in various populations. Moreover, a recent randomized controlled trial during spine surgery in adults has found ANIi to decrease the intraoperative and postoperative opioid consumption when used intraoperatively for guiding the administration of opioid agents

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years at time of surgery;
* Surgical correction of idiopathic scoliosis with or without thoracoplasty;
* Weight ≥ 30 kg : in order to allow using target plasma concentration administration of the opioid (remifentanil) and anaesthetic (propofol) agents; (pharmacokinetics models are not validated under this weight) during the intraoperative period;
* ASA (American Society of Anesthesiologist) status I to III
* Affiliation to the French national health insurance

Exclusion Criteria:

* Second time of a scoliosis correction in the preceding year (apart the use of halo-gravity traction or non-painful procedures such as digestive endoscopy);
* Chronic treatment (> 3 months) with: opioid agents, anti-epileptic agents or anti-depressant agents;
* Bad French language understanding;
* Expected difficulties in self-managing pain using the patient-controlled analgesia devices;
* ASA (American Society of Anesthesiologist) status IV or V;
* Any contraindication to one of the compound of the study: propofol, remifentanil, atracurium, paracetamol, Non-steroidal anti-inflammatory agents.
* Patients with a heart pace-maker device
* Patient under anti-arrythmic treatment

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
to evaluate the cumulative dose (in mg) of morphine during the first postoperative 24 hours according to the use or not of the ANI monitor (ANIi parameter) for guiding intraoperative opioid administration. | 24 hours
  Cumulative dose of morphine in first 24hrs post-operator

CONTACTS AND LOCATIONS:
Overall Officials: Souhayl Dahmani, MD-PhD, Principal Investigator — APHP
Locations (1):
- Department of Anesthesiology, Robert Debre University Hospital, Paris, France